CLINICAL TRIAL: NCT02300558
Title: A Phase 3, Single-Blind Study to Evaluate the Effect of Eleclazine (GS-6615) on Shortening of the QT Interval, Safety, and Tolerability in Subjects With Long QT Syndrome Type 3
Brief Title: Effect of Eleclazine on Shortening of the QT Interval, Safety, and Tolerability in Adults With Long QT Syndrome Type 3
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: GS-US-372-1234; 2014-000042-30 (EudraCT Number)
Record Dates: First submitted 2014-11-21; First posted 2014-11-25 (Estimated); Results first posted 2018-01-12 (Actual); Last update posted 2018-01-12 (Actual); Status verified 2017-12

CONDITIONS: Long QT Syndrome Type 3
Keywords: Type 3 long QT syndrome (LQT3); Long QT syndrome; Congenital long QT; Sudden cardiac death
MeSH Terms: conditions — Long QT syndrome type 3; Long QT Syndrome; Death, Sudden, Cardiac | interventions — eleclazine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Eleclazine (Single-blind treatment phase) (Experimental): Eleclazine and/or eleclazine placebo up to Week 24
  Interventions: Drug: Eleclazine; Drug: Eleclazine placebo
- Open-label Extension Phase (Experimental): Eligible participants will continue to receive open-label eleclazine until this drug is commercially available for the treatment of patients with LQT3, or until Gilead terminates development of eleclazine for the treatment of patients with LQT3, or the investigator deems it no longer in the participant's best interest.
  Interventions: Drug: Eleclazine

INTERVENTIONS:
Drug: Eleclazine — Tablets administered orally
  Other Names: GS-6615
Drug: Eleclazine placebo — Tablets administered orally
  Arms: Eleclazine (Single-blind treatment phase)

SUMMARY:
The primary objective of this study is to evaluate the effect of oral eleclazine on mean daytime QTcF interval after 24 weeks of treatment with elecalzine in participants with long QT syndrome Type 3. During the single-blind treatment period (24 weeks), participants will receive eleclazine and/or eleclazine placebo. Following the single-blind treatment period, participants who have not permanently discontinued study drug will be eligible, at the discretion of the investigator, to continue receiving eleclazine during an open-label extension (OLE) phase.

ELIGIBILITY:
Key Inclusion Criteria:

* Individuals with an established diagnosis of LQT3 (by genotype testing)
* Mean (of triplicate) QTc interval ≥ 480 msec (or ≥ 460 msec, for individuals who are currently taking ranolazine or Class I antiarrhythmic drugs such as mexiletine) at 3 or more time points, determined by standard 12-lead ECG, at screening

Key Exclusion Criteria:

* Known mutations associated with type 1 long QT syndrome (LQT1) or type 2 long QT syndrome (LQT2)
* Known or suspected history of seizures or epilepsy
* History of heart failure defined as New York Heart Association (NYHA) Class IV and/or known left ventricular ejection fraction (EF) ≤ 45%
* Body mass index (BMI) ≥ 40 kg/m^2 at screening
* Severe renal impairment at screening (defined as an estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73m^2, using the 4 Variable Modification of Diet in Renal Disease (MDRD) equation, as determined by the study center)
* Abnormal liver function tests at screening, defined as alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2 x upper limit of normal (ULN), or total bilirubin > 1.5 x ULN
* An aborted cardiac arrest (ACA), implantable cardioverter-defibrillator (ICD) implantation, syncopal episode, or appropriate ICD therapy within 3 months prior to screening
* Any other condition or circumstance that in the opinion of the investigator would preclude compliance with the study protocol

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2014-12-17 (Actual); Primary Completion 2016-12-12 (Actual); Study Completion 2017-02-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (12):
- United States (3):
  - Mayo Clinic Rochester, Rochester, Minnesota
  - NYU Langone Medical Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
- Nova Scotia Health Authority, Halifax, Nova Scotia, Canada
- France (3):
  - L'institut Du Thorax Nantes, Nantes
  - Groupe Hospitalier Bichat Claude Bernard, Paris
  - CHU Réunion Sud, Saint-Pierre
- LMU Klinikum der Universität München, München, Germany
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel
- Fondazione Salvatore Maugeri IRCCS, Pavia, Italy
- Academisch Medisch Centrum Amsterdam, Amsterdam, Netherlands
- Barts and The London School of Medicine and Dentistry, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in North America, Europe, and Asia. The first participant was screened on 17 December 2014. The last study visit occurred on 15 February 2017.
Pre-assignment Details: 54 participants were screened.
Groups:
- Eleclazine: * Single-Blind Treatment Period: Single oral loading dose of placebo to match eleclazine loading dose (8 x 6 mg placebo to match tablets) on Day 1; eleclazine 48 mg ( 8 x 6 mg tablets) on Day 2; followed by eleclazine 3 mg (1 x 3 mg tablet) once daily from Day 3 to the Week 12 Visit; then once daily maintenance dose of eleclazine 6 mg (1 x 6 mg tablet) from the day after the Week 12 Visit through Week 24
  * Open-label Extension (OLE): Eleclazine 6 mg or 3 mg tablets orally once daily
Period: Single Blind Phase (24 Weeks)
Arm/Group | Eleclazine
Started | 41
Completed | 35
Not Completed | 6
Not completed — Study Terminated by Sponsor | 6
Period: Open-Label (OL) Extension Phase
Arm/Group | Eleclazine
Started (3 participants completed the single-blind phase (24 weeks) but did not continue to OL Extension.) | 32
Completed | 0
Not Completed | 32
Not completed — Lack of Efficacy | 2
Not completed — Withdrew Consent | 1
Not completed — Study Terminated by Sponsor | 29

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: participants who received at least 1 dose of study drug (either active or placebo).
Groups:
- Eleclazine: * Single-Blind Treatment Period: Single oral loading dose of placebo to match eleclazine loading dose (8 x 6 mg placebo to match tablets) on Day 1; eleclazine 48 mg ( 8 x 6 mg tablets) on Day 2; followed by eleclazine 3 mg (1 x 3 mg tablet) once daily from Day 3 to the Week 12 Visit; then once daily maintenance dose of eleclazine 6 mg (1 x 6 mg tablet) from the day after the Week 12 Visit through Week 24
  * OLE: Eleclazine 6 mg or 3 mg tablets orally once daily
Arm/Group | Eleclazine
Number analyzed (Participants) | 41
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 17
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Black or African American | 0
  Native Hawaiian or Other Pacific Islander | 0
  White | 36
  Not Permitted | 1
  Other | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 40
  Not Permitted | 1
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 1
  Netherlands | 3
  United States | 11
  Italy | 12
  United Kingdom | 1
  Israel | 3
  France | 9
  Germany | 1
Mean Daytime QTcF Lead V5 (Standard 12-lead ECG) [Mean (Standard Deviation); unit: msec] — * QTcF refers to QT interval corrected for heart rate using the Fridericia formula. QTcF = QT/cube root (RR), where RR is in seconds.
  * AUC0-6 for QTcF was calculated using the trapezoidal rule, mean of triplicate values, and actual time (latest of triplicate times).
  * Mean daytime QTcF (AUC0-6/6) was computed by dividing AUC0-6 by the time from dosing to the 6 hour postdose time point.
  msec | 507.5 (38.11)
Mean Daily QTcF in Lead V5 (Holter) [Mean (Standard Deviation); unit: msec] — * AUC (0-6) was calculated using the trapezoidal rule, mean of triplicate vales, and nominal time.
  * Mean daytime QTcF (AUC 0-6/6) was computed by dividing AUC(0-6) by the time from the first nonmissing time^ to the last nonmissing time^, from predose to 6 hours postdose.
  * Mean nocturnal QTcF (AUC 0-6/6) was computed by dividing AUC(0-6) by the time from the first nonmissing time^ to the last nonmissing time^, from midnight to 6:00 AM.
  * Daily was computed as the average of daytime AUC(0-6/6) and nocturnal AUC (0-6/6), when both values are not missing.
  * ^ = nominal time point
  msec | 514.7 (45.76)
Mean Nocturnal QTcF in Lead V5 (Holter) [Mean (Standard Deviation); unit: msec] — AUC(0-6) for QTcF was calculated using the trapezoidal rule, mean of triplicate values, and nominal time.
  Mean nocturnal QTcF (AUC 0-6/6) was computed by dividing AUC(0-6) by the time from the first nonmissing nominal time point to the last nonmissing nominal time point, from midnight to 6:00 AM.
  msec | 530.6 (52.25)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Daytime QT Interval in Lead V5 Corrected for Heart Rate Using the Fridericia Formula (QTcF) Interval to Week 24 (Based on Standard 12-lead ECG Data)
Description: * Baseline was the Day 1 value.
  * QTcF is corrected QT interval using Fridericia's formula. QTcF = QT/cube root (RR), where RR is in seconds.
  * AUC0-6 for QTcF was calculated using the trapezoidal rule, mean of triplicate values, and actual time (latest of triplicate times).
  * Mean daytime QTcF (AUC0-6/6) was computed by dividing AUC0-6 by the time from dosing to the 6 hour postdose time point.
Time Frame: Baseline; Week 24
Population: Participants in Full Analysis Set (FAS) with available data were analyzed. FAS was defined as all enrolled participants who have confirmed LQT3 genotype, do not have confirmed LQT1 or LQT2 mutations, received at least 1 dose of active eleclazine, and have both a baseline and at least 1 postbaseline mean daytime QTcF interval (standard 12-lead).
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Eleclazine
Number analyzed (Participants) | 35
msec | -8.5 (18.03)
Statistical Analysis 1: Comparison: Eleclazine; Based on a 2-sided, paired t-test ( α = 0.05), and a standard deviation (SD) of 30 msec, a sample size of 40 participants provided greater than 95% power assuming a difference in mean daytime QTcF interval (AUC0-6/6) as measured by standard 12-lead ECG between baseline and Week 24 of 20 msec. The null hypothesis was that the mean difference between the baseline and Week 24 mean daytime QTcF interval was zero; Test type: Other; p = 0.0087, paired t- test

2. Secondary Outcome: Change From Baseline in Mean Daytime QTcF Interval (AUC0-6/6) to Week 12 (Lead V5; Standard 12-lead ECG)
Description: * Baseline was the Day 1 value.
  * QTcF is corrected QT interval using Fridericia's formula. QTcF = QT/cube root (RR), where RR is in seconds.
  * AUC0-6 for QTcF was calculated using the trapezoidal rule, mean of triplicate values, and actual time (latest of triplicate times) .
  * Mean daytime QTcF (AUC0-6/6) was computed by dividing AUC0-6 by the time from dosing to the 6 hour postdose time point.
Time Frame: Baseline; Week 12
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (95% Confidence Interval); unit: msec
Arm/Group | Eleclazine
Number analyzed (Participants) | 40
msec | 2.2 [-4.7 to 9.2]

3. Secondary Outcome: Change From Baseline in Mean Daily (Daytime and Nocturnal) QTcF Interval to Week 24 (Lead V5; Holter)
Description: * Baseline was the Day 1 value.
  * QTcF is corrected QT interval using Fridericia's formula. QTcF = QT/cube root (RR), where RR is in seconds.
  * Mean daytime QTcF (AUC0-6/6) was computed by dividing AUC0-6 by the time from the first nonmissing nominal time point to the last nonmissing nominal time point, from predose to 6 hours postdose. Mean nocturnal QTcF (AUC0-6/6) was computed by dividing AUC0-6 by the time from the first nonmissing nominal time point to the last nonmissing nominal time point, from midnight to 6:00 AM. Daily was computed as the average of daytime (AUC0-6/6) and nocturnal (AUC0-6/6), with both values required to compute the average.
Time Frame: Baseline; Week 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (95% Confidence Interval); unit: msec
Arm/Group | Eleclazine
Number analyzed (Participants) | 30
msec | -1.8 [-13.6 to 10.0]

4. Secondary Outcome: Change From Baseline in Mean Nocturnal QTcF Interval to Week 24 (Lead V5; Holter)
Description: * Baseline was the Day 1 value.
  * QTcF is corrected QT interval using Fridericia's formula. QTcF = QT/cube root (RR), where RR is in seconds.
  * Mean nocturnal QTcF (AUC0-6/6) was computed by dividing AUC0-6 by the time from the first nonmissing nominal time point to the last nonmissing nominal time point, from midnight to 6:00 AM.
Time Frame: Baseline; Week 24
Population: Participants in the the Full Analysis Set with available data were analyzed.
Measure: Mean (95% Confidence Interval); unit: msec
Arm/Group | Eleclazine
Number analyzed (Participants) | 31
msec | -3.0 [-17.1 to 11.0]

ADVERSE EVENTS:
Time Frame: Day 1 to the last dose date plus 30 days (median exposure to eleclazine: 396 days)
Description: Safety Analysis Set
Groups:
- Placebo: Single oral loading dose of placebo to match eleclazine loading dose (8 x 6 mg placebo to match tablets) on Day 1
- Eleclazine Loading Dose (LD) 48 mg: Eleclazine 48 mg ( 8 x 6 mg tablets) administered orally on Day 2
- Eleclazine Maintenance Dose (MD) 3 mg: Eleclazine 3 mg (1 x 3 mg tablet) administered once daily from Day 3 to the Week 12 Visit
- Eleclazine MD 6 mg: Eleclazine 6 mg (1 x 6 mg tablet) administered orally from the day after the Week 12 Visit through Week 24 and open-label extension.
- All Eleclazine: * Loading Dose: Eleclazine 48 mg ( 8 x 6 mg tablets) administered on Day 2 and 3 mg (1 x 3 mg tablet) once daily from Day 3 to the Week 12 Visit
  * Maintenance dose: Eleclazine 6 mg (1 x 6 mg tablet) from the day after the Week 12 Visit through Week 24 and open-label extension.
  Adverse events in this reporting group include those that occurred any time during the study by participants while receiving loading dose or maintenance dose of eleclazine.
Arm/Group | Placebo | Eleclazine Loading Dose (LD) 48 mg | Eleclazine Maintenance Dose (MD) 3 mg | Eleclazine MD 6 mg | All Eleclazine
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/41 | 0/41 | 0/41 | 0/41
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/41 | 1/41 | 0/41 | 1/41
Other Adverse Events (participants affected / at risk) | 5/41 | 5/41 | 17/41 | 14/41 | 24/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=41) | Eleclazine Loading Dose (LD) 48 mg (N=41) | Eleclazine Maintenance Dose (MD) 3 mg (N=41) | Eleclazine MD 6 mg (N=41) | All Eleclazine (N=41)
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=41) | Eleclazine Loading Dose (LD) 48 mg (N=41) | Eleclazine Maintenance Dose (MD) 3 mg (N=41) | Eleclazine MD 6 mg (N=41) | All Eleclazine (N=41)
Vertigo (Ear and labyrinth disorders) | 1 | 2 | 0 | 2 | 3
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 3 | 1 | 4
Nausea (Gastrointestinal disorders) | 0 | 1 | 3 | 0 | 4
Asthenia (General disorders) | 1 | 0 | 2 | 1 | 3
Fatigue (General disorders) | 0 | 0 | 3 | 2 | 5
Influenza (Infections and infestations) | 0 | 0 | 3 | 3 | 6
Nasopharyngitis (Infections and infestations) | 0 | 0 | 2 | 2 | 4
Weight increased (Investigations) | 0 | 0 | 1 | 2 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 2 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 0 | 3
Dizziness (Nervous system disorders) | 0 | 2 | 2 | 0 | 4
Headache (Nervous system disorders) | 2 | 1 | 2 | 4 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years